CLINICAL TRIAL: NCT01760876
Title: Evaluation of Healing the Biofreedom Stent Study
Brief Title: Evaluation of HealinG of Polymer-Free Biomlimus A9-Coated Stent by Optical Coherence Tomography (EGO-BIOFREEDOM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Stephen Lee (Other)
Responsible Party: Sponsor-Investigator, Professor Stephen Lee, Professor and Chief, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 12-454
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Coronary Disease
Keywords: Optical Coherence Tomography; Biofreedom Stent
MeSH Terms: conditions — Coronary Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biofreedom stent (Experimental): Coronary intervention
  Interventions: Device: coronary intervention

INTERVENTIONS:
Device: coronary intervention — The BioFreedom drug coated stent (DCS) Coronary Stent Delivery System is comprised of three key components

SUMMARY:
Since polymers have been identified as a possible cause of late complications of drug eluting stents, new stents are being designed to improve polymers' biocompatibility or to bond drugs on stents without polymers.

Biolimus A9 is the therapeutic agent used in the BioFreedom drug coated stent. Biolimus A9 is a proprietary semi-synthetic sirolimus derivative. It is highly lipophilic, rapidly absorbed in tissues, and able to reversibly inhibit growth factor-stimulated cell proliferation.

In this study, we use intracoronary optical coherence tomography (OCT) to evaluate the BioFreedom Stents after implantation regarding endovascular healing over time as primary objective; and also to evaluate secondary OCT, angiographic and clinical outcomes at various specific time points.

DETAILED DESCRIPTION:
Intra-coronary stenting is currently the standard of care post-balloon angioplasty for ischemic heart disease. Traditionally, bare metal stent (BMS) is used but in recent years it has been largely been replaced by drug-eluting stent (DES) which has reduced rates of restenosis. (1) However, the long term safety of DES still remains controversial due to reports of late stent thrombosis which presumably occurs secondary to delayed arterial healing and local hypersensitivity reactions which may be related to the drug, the polymer, or both. (2). Virmani et al (3) reported that patients who died of late stent thrombosis 18 months after sirolimus-eluting stent (SES) implantation showed a severe localized hypersensitivity reaction that involved the whole vessel wall and this reaction may be caused by polymer or from the drug-release kinetics of SES. It is known from preclinical and clinical studies that, nonabsorbable polymer can induce persistent inflammation which may lead to delayed cellular proliferation and 'late catch-up' restenosis (4).

Early (ie first) generation DES consisted of a metal stent for vessel scaffolding, cytotoxic drug for neointimal growth inhibition and a polymer coating to improve the biocompatibility of the stents or as a vehicle to load drugs onto stents. Since polymers have been identified as a possible cause of late complications of DES, new stents are being designed to improve polymers' biocompatibility or to bond drugs on stents without polymers. Biodegradable polymers are likely to be safer than nonabsorbable polymers because inflammation will be eliminated after the polymer degrades.

The BioFreedom drug coated stent (DCS) Coronary Stent Delivery System is comprised of three key components including 1) a 316 L stainless steel bare metal stent platform which has been modified with a proprietary surface treatment resulting in a selectively micro-structured, abluminal surface. The selectively micro-structured surface allows 2) Biolimus A9TM (drug) adhesion to the abluminal surface of the stent without the use of a polymer or binder. The drug-coated stent is crimped onto 3) a delivery system which includes a high pressure, semi-compliant balloon incorporated onto the distal tip of a rapid exchange delivery catheter system. The delivery system has two radiopaque markers inside the balloon, which fluoroscopically mark the ends of the stent to facilitate proper stent placement.

Biolimus A9 is the therapeutic agent used in the BioFreedom DCS. Biolimus A9 is a proprietary semi-synthetic sirolimus derivative. It is highly lipophilic, rapidly absorbed in tissues, and able to reversibly inhibit growth factor-stimulated cell proliferation. Current data suggest that Biolimus A9, on a molecular level, forms a complex with the cytoplasmic proteins that inhibit the cell cycle between the G0 and G1 phase. The result is an interruption of the cascade governing cell reproduction, growth, and proliferation. Related pharmaceuticals, sirolimus and everolimus, are well tolerated cytostatic immunosuppressive agents with predictable and similar adverse event profiles. Biolimus A9 is closely related chemically to both sirolimus and everolimus. Based on administration in healthy volunteers, Biolimus A9 has been shown to have a very similar adverse event profile to these other two drugs when used at equivalent dose levels., Biolimus A9 easily crosses the cell membrane to achieve therapeutic effects in target smooth muscle cells and, compared with the sirolimus-eluting Cypher stent (SES), the high lipophilicity of BA9 leads to relatively low systemic exposure.(5) Furthermore, the drug coating is applied only to the abluminal surface of the stent, allowing the drug release to be directed almost entirely into the vessel wall where it targets the smooth muscle cells injured by the angioplasty procedure. On the other hand, there is little drug release on the luminal surfaces of the stent, thus there is less inhibition of endothelial cells which need to grow on the inside of the stent in order for healing to occur.

Animal studies have shown the Biofreedom stent demonstrates equivalent or less early and late reduction of intimal smooth muscle cell proliferation compared with the Cypher Sirolimus-eluting stent (SES) in a porcine model. After implantation of BioFreedom stent, delayed arterial healing has been shown to be minimal, and there was no increased inflammation at 180 days compared with SES implantation (6). Pharmacokinetic and tissue concentration analyses showed that there was no high early peaking of Biolimus A9 level in blood (6). On-going studies of Biofreedom in humans showed non-inferiority of in-stent late lumen loss at 12 months versus paclitaxel eluting stents (PES) (7).

This current EGO BIOFREEDOM study protocol is designed based on the approved protocols of the EGO Study and EGO-COMBO Study, which were both successfully completed. We aim to focus mainly on the time frame, degree of endothelialization, and the subsequent neointimal proliferation after BioFreedom stent implantation, as assessed by the state-of-the-art intracoronary imaging - optical coherence tomography (OCT), which has been used extensively in the completed EGO and EGO-COMBO study.

Indeed, intracoronary optical coherence tomography (OCT) is a simple catheter-based imaging technique using optic fibre to achieve very detailed assessment (resolution down to 100 microns) in intra-coronary stent apposition, early stent coverage (endothelialization) and late stent neoinitmal growth (restenosis). It is performed as part of routine cardiac catheterization procedure and provides high-resolution cross sectional images of the coronary arteries. OCT has been shown to be safe in clinical practice (8). The LightLab C7XR OCT system (Frequency Domain OCT) is a commercial available product with CE Mark and FDA approval, which has been used in the EGO Studies. The OCT catheter is a non-occlusive optic fibre which is extremely small and flexible. It poses no additional risk to the patient other than those inherent risks of a standard angioplasty procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-85 years old
* Patient indicated for percutaneous coronary intervention with coronary artery disease and without contraindications to implantation of drug eluting stents
* Patient who agrees to have follow-up coronary angiograms

Exclusion Criteria:

* Patient who refuses to consent to multiple coronary angiograms or coronary angioplasty

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen WL Lee, MD FRCP FACC, Principal Investigator — Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hospital Authority
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hospital Authority, Hong Kong, Hong Kong

REFERENCES:
- [Result] Sousa JE, Costa MA, Abizaid AC, Rensing BJ, Abizaid AS, Tanajura LF, Kozuma K, Van Langenhove G, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Sustained suppression of neointimal proliferation by sirolimus-eluting stents: one-year angiographic and intravascular ultrasound follow-up. Circulation. 2001 Oct 23;104(17):2007-11. doi: 10.1161/hc4201.098056. PMID 11673337
- [Result] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Result] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Result] Kornowski R, Hong MK, Tio FO, Bramwell O, Wu H, Leon MB. In-stent restenosis: contributions of inflammatory responses and arterial injury to neointimal hyperplasia. J Am Coll Cardiol. 1998 Jan;31(1):224-30. doi: 10.1016/s0735-1097(97)00450-6. PMID 9426044
- [Result] Ostojic M, Sagic D, Jung R, Zhang YL, Nedeljkovic M, Mangovski L, Stojkovic S, Debeljacki D, Colic M, Beleslin B, Milosavljevic B, Orlic D, Topic D, Karanovic N, Paunovic D, Christians U; NOBORI PK Investigators. The pharmacokinetics of Biolimus A9 after elution from the Nobori stent in patients with coronary artery disease: the NOBORI PK study. Catheter Cardiovasc Interv. 2008 Dec 1;72(7):901-8. doi: 10.1002/ccd.21775. PMID 19016466
- [Result] Tada N, Virmani R, Grant G, Bartlett L, Black A, Clavijo C, Christians U, Betts R, Savage D, Su SH, Shulze J, Kar S. Polymer-free biolimus a9-coated stent demonstrates more sustained intimal inhibition, improved healing, and reduced inflammation compared with a polymer-coated sirolimus-eluting cypher stent in a porcine model. Circ Cardiovasc Interv. 2010 Apr;3(2):174-83. doi: 10.1161/CIRCINTERVENTIONS.109.877522. PMID 20407114
- [Result] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From Dec 20, 2012 to July 24, 2014, 106 patients enrolled for BioFreedom stent implantation and agreed to participate in the study at Queen Mary Hospital, Hong Kong.
Pre-assignment Details: 100 patients should be enrolled and randomly assigned to 5 monthly groups (n = 20:20:20:20:20) but 6 patients could not complete all the 3 OCT assessments (0 to 9 months) for reasons stated below and therefore a total of 106 patients were enrolled with BioFreedom study stents implanted and agreed for the study.
Groups:
- Biofreedom Stent: Coronary intervention: The BioFreedom drug coated study stent (DCS) is a polymer-free biolimus A9 coated drug stent. 100 patients needed to complete 3 OCT assessments over 9 months:- (1) at baseline (n = 100) for best stent optimization, (2) at 5 monthly groups (randomly assigned in 1 to 5 months n= 20:20:20:20:20) for early healing profile, and (3) at 9 months (n = 100) for neointima metrics.
Period: Overall Study
Arm/Group | Biofreedom Stent
Started | 106
Completed | 100 (12 months clinical FU of last patient in July 2015.)
Not Completed | 6
Not completed — Non-cardiac death (head injury) | 1
Not completed — Carcinoma of prostate | 1
Not completed — Impaired renal function | 1
Not completed — Major depression | 1
Not completed — Very poor baseline OCT quality | 2

BASELINE CHARACTERISTICS:
Population: All patients with coronary disease requiring stent implantation (BioFreedom) stent with (1)successful (evaluable) baseline OCT obtained, (2) 1 to 5 months 2nd OCT follow-up, and (3) 9 months 3rd OCT follow-up. 4 patients withdrew (1 renal failure, 1 emotionally unstable,1 died from fall and 1 withdrew due to personal reasons).
Groups:
- Biofreedom Stent: Coronary intervention: The BioFreedom drug coated study stent (DCS) is a polymer-free abluminally coated Biolimus A9 coated drug stent. 100 patients needed to complete 3 OCT assessments over 9 months:- (1) at baseline (n = 100) for best stent optimization, (2) at 5 monthly groups (randomly assigned in 1 to 5 months n= 20:20:20:20:20) for early healing profile, and (3) at 9 months (n = 100) for neointima metrics.
Arm/Group | Biofreedom Stent
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.99 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 89
Region of Enrollment [Number; unit: participants]
  Hong Kong | 104

OUTCOME MEASURES:

1. Primary Outcome: OCT Findings on Coverage (Degree of Endothelialisation/Coverage) From 1 to 9 Months.
Description: The percentage of strut coverage and category of coverage (A to F) from 1 month to 9 months by longitudinal sequential OCT assessments.
  A. Definitely uncovered - strut not covered by tissue, and both sides appear square; B. Uncovered with abnormal in-stent tissue - strut covered by irregular tissue or fibrin, and both sides appear square; C. Partially uncovered - strut partially covered by tissue but only one side has a smooth continuous shoulder; D. Covered (protruding) - strut covered by thin continuous tissue on both sides but still extending into the lumen; E. Covered (embedded) - strut covered by continuous tissue or neointima and not interrupting the smooth lumen contour; F. Covered (proliferative) - strut covered with excessive growth of neointima with thickness >0.3 mm.
Time Frame: 1 to 9 months
Population: 100 patients treated with BF stents and randomly assigned to 5 monthly groups (n = 20:20:20:20:20) at 1 to 5 months receiving OCT follow-up, and then 100 patients altogether at 9 months for another follow-up.
Measure: Median (Inter-Quartile Range); unit: percentage of strut coverage (D+E+F)
Groups:
- Biofreedom Stent: The healing profile (curve) in terms of percentage strut coverage of the BioFreedom Stent increased from a median of 85.77%, 86.95%, 88.56%, 96.79%, and 97.14% in the first 5 months, to 99.55% at 9 months.
Arm/Group | Biofreedom Stent
Number analyzed (Participants) | 100
percentage of strut coverage (D+E+F)
  1 Month (n=20) | 85.77 [79.1 to 90.25]
  2 Month (n=20) | 86.95 [81.55 to 94.44]
  3 Month (n=20) | 88.56 [84.62 to 97.63]
  4 Month (n=20) | 96.79 [94.31 to 98.7]
  5 Month (n=20) | 97.14 [95.31 to 99.01]
  9 Month (n=100) | 99.55 [98.17 to 99.93]

2. Secondary Outcome: OCT Endpoints (Neointimal Metrics), QCA Endpoints (Late Lumen Loss at 9 Months), and Clinical Endpoints (MACE at 9 Months and 12 Months). A Subgroup Analysis Would be Performed for Diabetic Patients.
Description: Secondary endpoints would consist of OCT endpoints (neointimal area, neointimal thickness, neointimal volume, and percentage neointimal volume ), QCA endpoints (late lumen loss at 9 months), and clinical endpoints (MACE, including stent thrombosis up to 12 months). A subgroup analysis will be performed for DM patients.
Time Frame: 9 months and 12 months
Reporting Status: Not Posted, anticipated posting 2017-12

ADVERSE EVENTS:
Time Frame: 1 year clinical follow up.
Description: 4 patients withdrew (1 renal failure, 1 emotionally unstable,1 died from fall and 1 withdrew due to personal reasons).
Groups:
- Biofreedom Stent: The BioFreedom drug coated study stent (DCS) is a polymer-free abluminally coated Biolimus A9 coated drug stent. 100 patients needed to complete 3 OCT assessments over 9 months:- (1) at baseline (n = 100) for best stent optimization, (2) at 5 monthly groups (randomly assigned in 1 to 5 months n= 20:20:20:20:20) for early healing profile, and (3) at 9 months (n = 100) for neointima metrics.
Arm/Group | Biofreedom Stent
Serious Adverse Events (participants affected / at risk) | 30/104
Other Adverse Events (participants affected / at risk) | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Biofreedom Stent (N=104)
Non-cardiac death from fall (Nervous system disorders) | 1/30 — Patient slipped and fell; admitted on 11 NOV 2013 with severe head injury (closed fracture of skill vault, cerebral contusion, subdural haematoma and subarachnoid hemorrhage). Patient died on 3 Dec 2013. (non-cardiac death - not related to MACE)
Admitted for "chest pain" in between 9 months (Cardiac disorders) | 2 — All 2 patients had no enzyme changes and no study-stent related ischaemia or infarct. All 2 patients discharged.
Admitted with left side numbness / stroke (Nervous system disorders) | 1 — Not cardiac related. MRI scheduled. Discharged.
Admitted for upper gastrointestinal bleeding (Gastrointestinal disorders) | 1 — Endoscopy performed. Treated and discharged.
Admitted for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 — No cause found. Discharged.
Admitted for chest infection (Respiratory, thoracic and mediastinal disorders) | 1 — Chest infection treated with antibiotics; all discharged.
Admitted for Colonoscopy (Gastrointestinal disorders) | 2 — Colonoscopy with polyps removed.
Admitted for epistaxis (Blood and lymphatic system disorders) | 1 — Treatment and discharged.
Admitted for epileptic attack (Nervous system disorders) | 1 — Treated and discharged.
Admitted for Hematoma at Vascular Femoral Access Site (Vascular disorders) | 1 — Anticoagulation and discharged.
Admitted for Acute Dermatitis (Reproductive system and breast disorders) | 1 — Admitted for penile and scrotal swelling. Treated by antibiotic and seen by surgeon. Discharged.
Admitted for low back pain (Musculoskeletal and connective tissue disorders) | 1 — Seen by orthopaedic surgeon and discharged.
Admitted for Acute Traumatic Closed Fracture of Left Foot (Musculoskeletal and connective tissue disorders) | 1 — Admitted for fractured bone (left calcaneum). Seen by orthopaedic surgeon and discharged.
Admitted for skin rashes, lower limb oedema (Renal and urinary disorders) | 1 — DM proteinuria in one patient. Two others mild oedema not having any overt heart failure. All discharged.
3 cases of in-stent restenosis at 9 months follow-up (Cardiac disorders) | 3 — 3 patients had in-stent restenosis of the BioFreedom study stent at 9 months follow-up and treated by another DES (RI). All discharged.
Admitted for Non-target Lesion Revascularization (Cardiac disorders) | 1 — Non-study lesion stented with BF stent shown ISR. Stented with ONYX.
Admitted For Atypical Chest Pain (Investigations) | 1 — Non-exertional. No evidence of disorders. Discharged.
Admitted For Fluid Retention (Renal and urinary disorders) | 1 — 24 hrs urine test done. Urine creatinine 2747, urine protein 5.48, Ur Prot/Ur Crea 346. Treated with ointment, diprosone oint. Skin condition improved
Admitted For Lower Leg Oedema (Renal and urinary disorders) | 1 — Provincial diagnosis: Nephrotic syndrome, possible charcot arthropathy. Increased ramipril 5mg bd, decreased metformin and fludrocortisone
Admitted For Palpitation (Investigations) | 1 — ECG revealed no ischemic changes. Physical examination and blood result were unremarkable. Blood pressure on high side was noted. Iosartan was increased to 25mg daily. Patient was stable and discharged home.
Admitted For Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 — The viral antigen detection (immunofluorescence) shown influenza B was positive.
Admitted For Urinary Tract Infection (Renal and urinary disorders) | 1 — Shortness of breath, cough, sputum, dizziness. Given augmentin IV. Discharged.
Admitted For NSTEMI (Cardiac disorders) | 1 — E admission on 14 Aug 2013 for chest pain. Trop. I 0.97ng/mL. Successful PCI to distal LM/ostial LAD lesion.
Admitted For Pyrexia of Unknown Origin (Investigations) | 1 — PET CT done and shown hypermetabolic para-aortoic LN. Blood culture and EMU for AFB negative. Impression was transient viral infection.
Admitted For Biliary Stone At Common Bile Duct (Hepatobiliary disorders) | 1 — The impression was post-cholecystectomy and CBD stone noted impacted at liver hilum by ultrasound. Patient was done the ERCP and found 3 large stones in the common duct. Discharged.

LIMITATIONS AND CAVEATS:
2 patients had difficult guiding-catheter engagement for optimal baseline OCT imaging with lots of blood-displacement artifacts; obtaining good future OCT assessments were impossible and were excluded from the study (replaced by another 2 patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No